CLINICAL TRIAL: NCT04162795
Title: An Open Label, Multi-center Study to Evaluate Sensory Attributes of an Antihistamine Product
Brief Title: A Study to Evaluate Cooling Sensation of an Allergy Product in Adults With a History of Allergies
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 21048
Record Dates: First submitted 2019-11-12; First posted 2019-11-14 (Actual); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Allergic Rhinitis
Keywords: Allergy; Upper respiratory allergies
MeSH Terms: conditions — Rhinitis, Allergic; Hypersensitivity | interventions — Loratadine

STUDY DESIGN:
Masking Description: Participants were blinded to product brand
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Loratadine chewable tablet (Experimental): Participants received one dose of loratadine chewable tablet to chew completely before swallowing.
  Interventions: Drug: Loratadine (Claritin, BAY76-2211)

INTERVENTIONS:
Drug: Loratadine (Claritin, BAY76-2211) — Chewable tablet, oral, single dose

SUMMARY:
In this study, researchers were primarily interested in evaluating the level of agreement of cooling sensation provided by this chewable, flavored, allergy medicine. Participants joining this study received one test drug tablet and were asked to chew completely before swallowing the drug. A questionnaire was used to collect the feedback from participants. The study involved only one (1) visit and participant stayed in this study for about 60-75 minutes to evaluate the cooling sensation as well as other sensory attributes perceived in the mouth, nose and throat.

ELIGIBILITY:
Inclusion Criteria:

* Female or male adults aged 18 to 65 years of age inclusive
* Were in good general health
* Previous self-reported sufferers of upper respiratory allergies who at the time of the study are either asymptomatic, symptomatic but not treating and agree to use study medication or symptomatic and treating with an allergy medicine that is not an antihistamine
* Agreed to not use antihistamine products 24 hours before and after the treatment
* Willing to avoid eating food or candy (other than crackers consumed during testing), drinking any liquid other than water, gum chewing and teeth brushing one hour prior to testing

Exclusion Criteria:

* Individuals who had used oral/systemic medications 24 hours before the first administration of test product
* Individuals who used medications which might influence taste perception
* Individuals who had received or used an investigational new drug in the last 30 days or had been an active participant in another clinical or market research study in the last 30 days
* Women who were pregnant or thinking of becoming pregnant or were nursing
* Participants with congestion at the time of study visit
* Any self-reported symptoms or conditions that might interfere with the participants ability to complete the evaluation of the product on testing day
* Any current medical condition that in the opinion of the Investigator or designee might interfere with normal taste and/or temperature perception (e.g., active common cold, sinus infection, bronchial infection, adenoids, paresthesia etc.)
* History of alcohol or drug abuse
* History of hypersensitivity or allergic reactions to any ingredients in the test product
* Individuals with a history of glaucoma, liver or kidney disease, respiratory conditions such as chronic bronchitis or swallowing difficulties
* Individuals who were currently wearing any kind of dental braces or with dental work or had cavities and associated pain that might affect their ability to chew a tablet

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 468 (Actual)
Dates: Start 2019-11-12 (Actual); Primary Completion 2019-11-13 (Actual); Study Completion 2019-11-13 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Focus Pointe Global, Teaneck, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided
Availability of this study's data will be determined according to Bayer's commitment to the EFPIA/PhRMA "Principles for responsible clinical trial data sharing". This pertains to scope, timepoint and process of data access. As such, Bayer commits to sharing upon request from qualified researchers patient-level clinical trial data, study-level clinical trial data, and protocols from clinical trials in patients for medicines and indications approved in the US and EU as necessary for conducting legitimate research. This applies to data on new medicines and indications that have been approved by the EU and US regulatory agencies on or after January 01, 2014. Interested researchers can use www.clinicalstudydatarequest.com to request access to anonymized patient-level data and supporting documents from clinical studies to conduct research. Information on the Bayer criteria for listing studies and other relevant information is provided in the Study sponsors section of the portal.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study was conducted at multiple centers in the US between 12 November 2019 (first participant first visit) and 13 November 2019 (last participant last visit).
Pre-assignment Details: Overall, 468 participants were screened. Of them, 10 participants were screen failures and 16 participants did not complete the study with early termination. 442 participants received study treatment and completed the study.
Period: Overall Study
Arm/Group | Loratadine Chewable Tablet
Started | 468
Completed | 442
Not Completed | 26
Not completed — Other | 16
Not completed — Screen failures | 10

BASELINE CHARACTERISTICS:
Population: All participants who received the study medication and had an evaluation data for study medication
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Age, Customized [Number; unit: Percentage of participants]
  18- 34 years | 30
  35- 44 years | 30
  45- 54 years | 26
  55+ years | 14
Sex/Gender, Customized [Number; unit: Percentage of participants]
  Male | 46
  Female | 54
Race/Ethnicity, Customized [Number; unit: Percentage of participants]
  White | 52
  Black/African American | 33
  Hispanic | 12
  Asian | 5
  Other races | 2

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Agreement of Perception of Cooling Sensation
Description: Participants were asked to response to question "the product provides a cooling sensation" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of perception of the sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.99 [0.98 to 1.00]

2. Secondary Outcome: Proportion of Participants With Agreement of Perception of Cooling Sensation Per Location
Description: Participants were asked to respond to question "the product provides a cooling sensation in the mouth, nose or throat" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of perception of the sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants
  Cooling in Mouth | 0.99 [0.98 to 1.00]
  Cooling in Nose | 0.71 [0.67 to 0.76]
  Cooling in Throat | 0.93 [0.90 to 0.95]

3. Secondary Outcome: Proportion of Participants With Agreement of Perception of Refreshing Sensation
Description: Participants were asked to response to question "the product provides a refreshing sensation" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of perception of the sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants
  Refreshing | 0.96 [0.94 to 0.98]
  ...Refreshing in Mouth | 0.96 [0.94 to 0.97]
  ...Refreshing in Nose | 0.61 [0.57 to 0.66]
  ...Refreshing in Throat | 0.88 [0.85 to 0.91]

4. Secondary Outcome: Proportion of Participants With Agreement of the Refreshing of the Cooling Sensation
Description: Participants were asked to response to question "the cooling sensation is refreshing" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of the refreshing of the cooling sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.96 [0.94 to 0.97]

5. Secondary Outcome: Proportion of Participants With Agreement of the Unique Sensory Experience for an Allergy Medicine
Description: Participants were asked to response to question "the sensory experience is unique for an allergy medicine" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of the unique sensory experience sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.94 [0.92 to 0.96]

6. Secondary Outcome: Proportion of Participants With Agreement of Soothing Feeling on the Throat
Description: Participants were asked to response to question "the product feels soothing on the throat" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of the soothing feeling.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.89 [0.86 to 0.92]

7. Secondary Outcome: Proportion of Participants With Agreement of Liking the Flavor Sensation of the Product
Description: Participants were asked to response to question "I like the flavor sensation of the product" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of liking the enjoyable flavor sensation.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.87 [0.83 to 0.90]

8. Secondary Outcome: Proportion of Participants With Agreement of the Enjoyable Product Experience
Description: Participants were asked to response to question "the product experience was enjoyable" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of the enjoyable experience.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.85 [0.81 to 0.88]

9. Secondary Outcome: Proportion of Participants With Agreement of the Great Taste of the Product
Description: Participants were asked to response to question "the product tastes great" using a 5 point agreement scale (range from 1=strongly disagree to 5=strongly agree). Selection of the top 2 choices (strongly agree and somewhat agree) from the scale was considered as agreement of the great taste.
Time Frame: Up to 5 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Number (95% Confidence Interval); unit: Proportion of participants
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Proportion of participants | 0.77 [0.73 to 0.81]

10. Secondary Outcome: Time to Perception of Cooling Sensation
Description: The mean time point at which cooling was initially perceived was claimed as the onset of cooling. The mean onsets of cooling sensation in the mouth, nose and throat were reported.
Time Frame: Up to 60 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Mean (95% Confidence Interval); unit: Seconds
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Seconds
  Cooling in Mouth: number analyzed (Participants) | 437
  Cooling in Mouth | 5.82 [5.33 to 6.32]
  Cooling in Nose: number analyzed (Participants) | 320
  Cooling in Nose | 14.97 [13.00 to 16.94]
  Cooling in Throat: number analyzed (Participants) | 410
  Cooling in Throat | 16.17 [14.43 to 17.91]

11. Secondary Outcome: Duration of Cooling Sensation
Description: Participants who reported that they never experienced a cooling sensation were not included in the model. Those for whom the cooling sensation extended for 60 minutes or more were considered right-censored and were treated as such in the model. The median time of cooling sensation in the mouth, nose and throat was reported. Dispersion values were not calculated for this sensory study.
Time Frame: Up to 60 minutes post ingestion of study medication
Population: All participants who received the study medication and had an evaluation data for study medication
Measure: Median (Full Range); unit: Minutes
Arm/Group | Loratadine Chewable Tablet
Number analyzed (Participants) | 442
Minutes
  Cooling in Mouth | 20 [NA to NA] — The analysis of duration of cooling sensation was based on a Kaplan-Meier survival model. The Kaplan-Meier figures are included in the study report but cannot be provided in this data set. The specific dispersion values are not included in the study report or source tables for this sensory study.
  Cooling in Nose | 20 [NA to NA] — The analysis of duration of cooling sensation was based on a Kaplan-Meier survival model. The Kaplan-Meier figures are included in the study report but cannot be provided in this data set. The specific dispersion values are not included in the study report or source tables for this sensory study.
  Cooling in the Throat | 15 [NA to NA] — The analysis of duration of cooling sensation was based on a Kaplan-Meier survival model. The Kaplan-Meier figures are included in the study report but cannot be provided in this data set. The specific dispersion values are not included in the study report or source tables for this sensory study.

ADVERSE EVENTS:
Time Frame: From the signing of the informed consent form (ICF) until discharge from the study site (1 day)
Arm/Group | Loratadine Chewable Tablet
All-Cause Mortality (participants affected / at risk) | 0/442
Serious Adverse Events (participants affected / at risk) | 0/442
Other Adverse Events (participants affected / at risk) | 9/442
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Loratadine Chewable Tablet (N=442)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Rhinitis (Infections and infestations) | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 2
Salivary duct inflammation (Gastrointestinal disorders) | 1
Dyspepsia (Gastrointestinal disorders) | 2
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Ocular sensory symptom (Eye disorders) | 1

LIMITATIONS AND CAVEATS:
Kaplan-Meier Estimates of the duration of the cooling sensation were not able to be reported in this data set.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-10-21): https://cdn.clinicaltrials.gov/large-docs/95/NCT04162795/Prot_SAP_000.pdf